CLINICAL TRIAL: NCT06642051
Title: Safety of the Sonablate System for the High-Intensity Focused Ultrasound (HIFU) Ablation of Incompetent Veins of the Periphery
Brief Title: Safety of the Sonablate HIFU System for the Ablation of Incompetent Veins of the Periphery
Acronym: HIFIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sonablate (Industry)
Collaborators: Vascular Care CT, PLLC (Other); Vascular Breakthroughs, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20243482
Record Dates: First submitted 2024-09-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Venous Insufficiency, CVI; Venous Malformations; Venous Leg Ulcers; Klippel-Trenaunay Syndrome; CLOVES Syndrome; Blue Rubber Bleb Nevus Syndrome
Keywords: High Intensity focused ultrasound; venous closure; endovenous ablation
MeSH Terms: conditions — Blindness, Cortical; Klippel-Trenaunay-Weber Syndrome; Congenital Lipomatous Overgrowth, Vascular Malformations, and Epidermal Nevi; Blue rubber bleb nevus syndrome

STUDY DESIGN:
Intervention Model Description: The use of High Intensity Focused Ultrasound for the ablation of incompetent veins of the periphery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Prospective observational (Experimental): Patients that have undergone high intensity focused ultrasound ablation of incompetent veins of the periphery
  Interventions: Device: High Intensity focused ultrasound

INTERVENTIONS:
Device: High Intensity focused ultrasound — Sonablate High Intensity Focused Ultrasound system to ablate incompetent veins of the periphery
  Other Names: Venous ablation

SUMMARY:
The goal of this clinical trial is to learn if the Sonablate High Intensity Focused Ultrasound device can be safely used to treat patients with Chronic Venous Incompetence (CVI) including those with venous malformations of the periphery meaning legs, abdomen, chest or back. Examples of CVI are varicose veins, vascular congestion, venous ulcer, venous clusters, venous anomalies, mixed malformation, Klippel-Trenaunay Syndrome, CLOVES, Syndrome, Blue Rubber bleb Nevus Syndrome. HIFU is a non-invasive treatment as opposed to current treatment options which include incisions, needle penetration, wire insertions or catheter insertions.

DETAILED DESCRIPTION:
The Sonablate High Intensity Focused Ultrasound (HIFU) system is a non-invasive technology that uses focused ultrasound waves to ablate targeted tissue within the body without ionizing radiation or surgical excision. Through the precise delivery of ultrasonic waves, HIFU rapidly elevates the temperature in the targeted tissue, leading to the disruption of lipid membranes, denaturation of proteins, destruction of vascular endothelial cells and ultimately coagulative necrosis without damage to the overlying tissue. This device is cleared by the FDA for the ablation of prostate tissue.

This is a single arm, single institution, Phase one trial of 30 patients planned to last 18 months. The primary endpoint is to assess the 30-day safety profile and technical feasibility of using the Sonablate high-intensity focused ultrasound (HIFU) system for ablating incompetent veins of the periphery. This includes vascular malformations, varicose veins and incompetent superficial veins.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of age 18 or older with clinical and imaging evidence of venous malformations and/or venous insufficiency of the periphery
2. Lesions no deeper than 4.0cm from the skin surface
3. Lesions appropriate for and patient amenable to HIFU therapy of targeted vascular lesion/structure as determined by the principal operator and investigator
4. Ability to provide treatment consent for Sonablate HIFU energy delivery
5. Ability and willingness to remain compliant with recommended post-op follow-up

Exclusion Criteria:

1. Patient unable or unwilling to provide consent
2. Patient unable or unwilling to undergo HIFU energy delivery
3. Patient with vascular lesions involving the central nervous system, face, head, and neck, genitalia, visceral or internal organs
4. Patient with known vasculitis or other inflammatory vasculopathies
5. Patients with active or prior history of DVT or PE
6. Any lesion deemed unsafe by the treating surgeon or PI of the study for HIFU at the time of treatment based on clinical assessment, ultrasonographic features and/or probe positioning limitations
7. Subject who has vascular tissue targets lying <1cm from sensitive structures or large vessels
8. Women who are pregnant or planning to become pregnant prior to procedure or within the 30-day study period, or nursing
9. Vulnerable patients
10. Subject with vessels >6 mm in diameter within the vascular tissue target

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety of Sonablate High-Intensity Focused Ultrasound probe for ablating incompetent veins of the periphery. | 30 days
  Safety as measured by the magnitude and frequency of adverse events from HIFU. This includes any burns, scalds, blistering and hyperemic changes on physical exam intraoperatively, at 6h, 24h, 1w, and 4 weeks post-operatively; worsening limb pain and swelling due to DVT diagnosed with Duplex Ultrasound within 4 weeks post-operatively; sensory nerve injury via formal neurological examination at 6h, 1w, and 4 weeks post-operatively.

SECONDARY OUTCOMES:
Short-term efficacy and technical feasibility of using the Sonablate High-Intensity Focused Ultrasound probe for ablating incompetent veins of the periphery | 30 days
  Real-time B mode ultrasound imaging of HIFU to vascular tissue to evaluate the ultrasonographic changes in the targeted vessels and immediately adjacent tissues. Intraoperative duplex ultrasound of the targeted veins to quantify vessel closure rates or thrombosis immediately after HIFU delivery. Post-operative duplex ultrasound or magnetic resonance imaging of the targeted veins during follow up at 1 week and 4 weeks to assess vessel closure rates or thrombosis of target veins.

CONTACTS AND LOCATIONS:
Overall Officials: Naiem Nassiri, MD, FSVS, RPVI, Principal Investigator — The Vascular Care Group
Locations (1):
- The Vascular Care Group, Darien, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vascular anomalies and malformation program patient information website — https://thevascularcaregroup.com/malformations/
- See also: Resource for information on vascular birthmarks, anomalies and related symptoms. — https://birthmark.org/
- See also: Comprehensive online information on the Sonablate high intensity focused ultrasound probe. — https://www.sonablate.com/
- See also: Comprehensive source of information for vast array of clinical applications for focused ultrasound therapy — https://www.fusfoundation.org/